CLINICAL TRIAL: NCT04790942
Title: Effect of Berberine Hydrochloride on Blood Pressure and Vascular Endothelial Function in Patients With Hypertension
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jun Tao (Other)
Responsible Party: Sponsor-Investigator, Jun Tao, Director, Head of the Department of Hypertension and Cardiovascular Disease, Principal Investigator, Clinical Professor, First Affiliated Hospital, Sun Yat-Sen University
Organization: First Affiliated Hospital, Sun Yat-Sen University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BBR-[2020]433
Record Dates: First submitted 2021-03-08; First posted 2021-03-10 (Actual); Last update posted 2021-03-10 (Actual); Status verified 2021-03

CONDITIONS: Hypertension; Endothelial Dysfunction; Blood Pressure
Keywords: berberine; hypertension; vascular endothelial function; brachial ankle pulse wave velocity; brachial artery blood flow-mediated vasodilation
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- berberine hydrochloride group (Experimental): the berberine hydrochloride group (BBR) take berberine hydrochloride tablets
  Interventions: Drug: berberine hydrochloride
- lifestyle intervention group (Placebo Comparator): Lifestyle intervention group (CON) refers to healthy lifestyle education
  Interventions: Behavioral: lifestyle intervention group

INTERVENTIONS:
Drug: berberine hydrochloride — the berberine hydrochloride group (BBR) take berberine hydrochloride tablets (0.4g, 3 times/day, 3 months)
  Other Names: BBR
  Arms: berberine hydrochloride group
Behavioral: lifestyle intervention group — The lifestyle intervention group (CON) mainly includes reducing sodium intake, healthy diet guidance, increasing exercise, quitting smoking and restricting alcohol consumption
  Other Names: CON
  Arms: lifestyle intervention group

SUMMARY:
Hypertension is a progressive cardiovascular syndrome caused by multiple causes, which can lead to changes in the function and structure of the heart and blood vessels. It is the leading risk factor of cardiovascular disease.

Berberine (BBR) hydrochloride is an isoquinoline alkaloid (chemical formula: C20H18NO4) extracted from traditional Chinese herb Coptis chinensis. It has been widely used to treat diarrhea and enteritis for hundreds of years in China. BBR has extremely high clinical application value. It is an over-the-counter drug with low price, good safety and few adverse reactions in China.

We found that Berberine (BBR) hydrochloride tablets have a hypotensive effect in clinical practice. However, there are few clinical studies on the treatment of hypertensive patients with BBR tablets. In addition, the clinical dosage of BBR tablets is not uniform, and its molecular mechanism is still unclear.

In order to further evaluate the clinical efficacy of BBR in reducing blood pressure and improving vascular endothelial injury, we carried out this clinical trial of drug intervention for hypertensive population.

After signed the informed consent, the subjects are assigned to the lifestyle intervention group (CON) and berberine hydrochloride group (BBR). The berberine hydrochloride group (BBR) take berberine hydrochloride tablets (0.4g, 3 times/day, 3 months) . We will follow up blood pressure and vascular endothelial function in 1 month and 3 months after taking the medicine.

ELIGIBILITY:
Inclusion Criteria:

1. Essential hypertension (office blood pressure: systolic blood pressure 140-159 mmHg and/or diastolic blood pressure 90-99 mmHg
2. 18 to 75 years old
3. No drugs or dietary supplements that affect blood pressure and vascular endothelial function have been used in the past 3 months, mainly including antihypertensive, lipid-lowering, hypoglycemic drugs and natural plant extract antioxidants
4. Individuals who voluntarily sign the consent form after being fully informed and understanding the purpose and procedure of the study, characters of the disease, drug effects, methods of related examinations, and potential risk/benefits of the study

Exclusion Criteria:

1. Individuals with secondary blood pressure rise factors
2. Individuals who are hypersensitive or intolerant to the drugs
3. Individuals presenting severe constipation
4. Individuals with severe heart disease, abnormal liver and kidney function, acute and chronic infections, autoimmune diseases and patients with any history of cancer
5. Individuals with mental diseases who are not able to cooperate
6. Pregnant women, women during breast-feeding period, or women with expect pregnancy
7. Individuals with hemolytic anemia and glucose-6 phosphate dehydrogenase deficiency

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-10-22 (Actual); Primary Completion 2022-02-22 (Estimated); Study Completion 2022-05-22 (Estimated)

PRIMARY OUTCOMES:
Office blood pressure | 3 months
  BP measurement was in accordance with the method recommended by clinical guidelines. After rest for at least 5 minutes, subjects were examined while seated in a quiet, temperature-controlled room, with the feet on the floor and arm supported at heart level. BP was measured using an automated device at least 2 measurements spaced 2 minutes apart, and additional measurements if the ﬁrst 2 are quite different. Average BP readings were recorded.
brachial-ankle pulse wave velocity (baPWV) | 3 months
  baPWV was measured by using an automatic device as reported previously and was expressed as centimeters per second (cm/sec). The measurement of baPWV is generally accepted as the simplest, robust, and reproducible method to represent arterial stiffness.

SECONDARY OUTCOMES:
24-hour ambulatory blood pressure monitoring (ABPM) | 3 months
  We record the 24 h ABPM results before recruitment and during the follow-up period.
brachial arterial flow-mediated dilation (FMD) | 3 months
  Subjects were recommended to rest for 10 min or longer and were examined in a quiet, temperature-controlled room. FMD was examined through noninvasive ultrasound scan; it could dynamically record artery diameter, at rest (baseline) and reactive hyperemia period produced by using the cuff inflated to the greater of 50 mmHg above systolic pressure or 200 mmHg for 5 min as previously described.

CONTACTS AND LOCATIONS:
Locations (1):
- Jun Tao, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No